CLINICAL TRIAL: NCT04180384
Title: A Safety Study of Oraxol (HM30181 + Oral Paclitaxel) in Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Athenex, Inc. (Industry)
Collaborators: Zenith Technology Corporation Limited (Industry); PharmaEssentia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KX-ORAX-003
Record Dates: First submitted 2019-06-13; First posted 2019-11-27 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: For 1 dosing week (at least 1 week following the paclitaxel capsule PK sampling period, ie, at Week 5 or later), a subgroup of 8 participants (Group B) will receive Oraxol as HM30181 plus a tablet formulation of paclitaxel. For the remainder of the study, Group B participants will receive the current clinical capsule formulation of paclitaxel. This will allow for comparison of the bioavailability of these 2 formulations with minimal impact on safety or activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oraxol (paclitaxel capsules+ HM30181AK-US) (Experimental): Oraxol paclitaxel - supplied as 30-mg capsules
  Oraxol HM30181 methansulfonate monohydrate - supplied as 15-mg HM30181AK-US tablets
  Interventions: Drug: Oraxol
- Oraxol (paclitaxel tablets+ HM30181AK-US) (Active Comparator): Oraxol paclitaxel - supplied as 30-mg tablets
  Oraxol HM30181 methansulfonate monohydrate - supplied as 15-mg HM30181AK-US tablets
  Interventions: Drug: Oraxol

INTERVENTIONS:
Drug: Oraxol — Paclitaxel:
  5β,20-Epoxy-1,2α,4,7β,10β,13α-hexahydroxytax-11-en-9-one 4,10-diacetate 2-benzoate 13- ester with (2R,3S)-N-benzoyl-3-phenylisoserine
  HM30181 methanesulfonate monohydrate:
  N-(2-(2-(4-(2-(6,7-Dimethoxy-3,4-dihydroisoquinolin-2(1H)-yl)ethyl)phenyl)-2H-tetrazol-5-yl)-4,5-dimethoxyphenyl)-4-oxo-4H-chromene-2-carboxamide Methanesulfonate monohydrate
  Other Names: HM30181 methanesulfonate monohydrate; Oral paclitaxel capsules; Oral paclitaxel tablets

SUMMARY:
Oraxol is a combination of an oral tablet, HM30181 methanesulfonate, and capsules that contain paclitaxel. HM30181 is a drug that helps the body absorb paclitaxel, a drug used to treat cancer. Initially this study is intended as an extension study of KX-ORAX-002 pharmacokinetic study for patients who wish to continue Oraxol treatment and who are eligible to participate. The purpose of this study is to check the safety and tolerability of Oraxol when it is administered on a weekly basis and to confirm the sustained oral bioavailability of paclitaxel following multiple dosing; also compare the relative bioavailability of paclitaxel tablets vs paclitaxel capsules (Group B only).

DETAILED DESCRIPTION:
Oraxol is a combination of an oral tablet, HM30181 methanesulfonate, and capsules that contain paclitaxel. HM30181 is a drug that helps the body absorb paclitaxel, a drug used to treat cancer. Initially this study is intended as an extension study of KX-ORAX-002 pharmacokinetic study for patients who wish to continue Oraxol treatment and who are eligible to participate. Once the dose of Oraxol has been confirmed in the KX-ORAX-002 study, then enrollment of patients who have not participated in the KX-ORAX-002 study can be allowed. The purpose of this study is to check the safety and tolerability of Oraxol when it is administered on a weekly basis and to confirm the sustained oral bioavailability of paclitaxel following multiple dosing; also compare the relative bioavailability of paclitaxel tablets vs paclitaxel capsules (Group B only). Participants in Group B (N=8) will receive the same weekly paclitaxel capsule treatment as the remainder of the subjects except for 1 dosing week (at least 1 week following the paclitaxel capsule PK sampling period) during which they will receive paclitaxel tablets and undergo PK assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Males and females ≥18 years of age on day of consent
3. Cancer patients for whom treatment with IV paclitaxel at 80 mg/m2 has been recommended by their oncologist, either as monotherapy or in combination with other agents
4. Adequate hematologic status:

   * Absolute neutrophil count (ANC) ≥1.5 x 10^9/L
   * Platelet count ≥100 x 10^9/L
   * Hemoglobin (Hgb) ≥90 g/L
5. Adequate liver function as demonstrated by:

   * Total bilirubin of ≤20 μmol/L or ≤30 μmol/L for participants with liver metastasis
   * Alanine aminotransferase (ALT) ≤3 x upper limit of normal (ULN) or ≤5 x ULN if liver metastasis is present
   * Alkaline phosphatase (ALP) ≤3 x ULN or ≤5 x ULN if liver or bone metastasis are present
   * ALP >5 x ULN if liver or bone metastasis are present and the major fraction of ALP is from bone metastasis, at the discretion of the Investigator
   * Gamma glutamyl transferase (GGT) <10 x ULN
6. Adequate renal function as demonstrated by serum creatinine ≤177 μmol/L or creatinine clearance >50 mL/min as calculated by the Cockcroft and Gault formula
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 16
8. Life expectancy of at least 3 months
9. Willing to fast for 8 hours before and 4 hours after Oraxol administration on all treatment days (but may have water 1 hour after completion of Oraxol dosing and as needed with other prescribed medications)
10. During the inpatient PK sampling week(s):

    * Willing to abstain from alcohol consumption for 3 days before the first dose of Oraxol through the completion of protocol-specified PK sampling for that treatment week
    * Willing to refrain from caffeine consumption for 12 hours before the first dose of Oraxol through the completion of protocol-specified PK sampling for that treatment week
11. Women must be postmenopausal (>12 months without menses) or surgically sterile (ie, by hysterectomy and/or bilateral oophorectomy) or, if of childbearing potential, must be using effective contraception (ie, oral contraceptives, intrauterine device, double barrier method of condom and spermicide) and agree to continue use of contraception for the duration of their participation in the study. Women of childbearing potential must agree to use contraception for 6 months after their last dose of study drug.
12. Sexually active male participants must use a barrier method of contraception during the study and agree to continue the use of male contraception for at least 6 months after the last dose of study drug.

Exclusion Criteria:

1. Currently taking a prohibited concomitant medication:

   * Strong inhibitors (eg, ketoconazole) or strong inducers (eg, rifampin or St. John's Wort) of cytochrome P450 (CYP) 3A4 (within 2 weeks prior to the start of dosing in the study)
   * Strong inhibitors (eg, gemfibrozil) or strong inducers (eg, rifampin) of CYP2C8 (within 2 weeks prior to the start of dosing in the study)
   * Strong P-gp inhibitors (eg, verapamil) or strong inducers (eg, rifampin). Participants who are taking such medications but who are otherwise eligible may be enrolled if they discontinue the medication ≥1 week before dosing and remain off that medication through the end of study treatment.
   * An oral medication with a narrow therapeutic index known to be a P-gp substrate (eg, digoxin, dabigatran) within 24 hours prior to start of dosing in the study
2. Use of warfarin. Participants receiving warfarin who are otherwise eligible and who may be appropriately managed with low molecular weight heparin, in the opinion of the Investigator, may be enrolled in the study provided they are switched to low molecular weight heparin at least 7 days prior to receiving study treatment.
3. Unresolved toxicity from prior chemotherapy (participants must have recovered all significant toxicity to ≤ Grade 1 CTCAE toxicity from previous anticancer treatments or previous investigational agents). This does not extend to symptoms or findings that are attributable to the underlying disease
4. Received investigational agents within 14 days or 5 half-lives prior to the first study dosing day, whichever is longer
5. Women of childbearing potential who are pregnant or breastfeeding
6. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, clinically significant myocardial infarction within the last 6 months, unstable angina pectoris, clinically significant cardiac arrhythmia, bleeding disorder, chronic pulmonary disease requiring oxygen, or psychiatric illness/social situations that would limit compliance with study requirements
7. Major surgery to the upper GI tract, or have a history of GI disease or other medical condition that, in the opinion of the Investigator may interfere with oral drug absorption
8. A known history of allergy to paclitaxel. Participants whose allergy was due to the IV solvent (such as Cremophor®) and not paclitaxel will be eligible for this study.
9. Any other condition which the Investigator believes would make a subject's participation in the study not acceptable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of Oraxol (Incidence of Treatment-Emergent Adverse Events) | From screening until final visit (within 28 days after the last dose of study drug was taken, and preferably before the participant receives any additional chemotherapy).
  Safety and tolerability as assessed by the incidence of adverse events. Treatment-emergent AEs (TEAEs) are defined as those AEs with an onset after dosing and those pre-existing AEs that worsen during the study.
  AEs will include those reported by participants as well as those observed by the clinical team, or clinically significant changes in lab tests, vital signs and ECGs. Possible AEs may include gastrointestinal effects and abdominal pain but as this is an early phase clinical trial and the likely AE profile is not yet known.

SECONDARY OUTCOMES:
Sustained oral bioavailability of paclitaxel following multiple dosing | PK samples will be collected during dosing for Week 4 or may be done during a later dosing week at the investigator's discretion and/or at the participant's convenience before patients' withdrawal from the study, up to 8 months.
  Oraxol PK data from this study will be compared with Oraxol PK data from study KX-ORAX-002.
the relative bioavailability of paclitaxel tablets vs paclitaxel capsules (Group B only) | PK samples will be collected during dosing for Week 5; or may be done during a later dosing week at the investigator's discretion and/or at the participant's convenience, up to 8 months.
  For Group B, 8 subjects will be enrolled and the geometric mean ratio (GMR) will be calculated comparing the Cmax and AUC0-∞ of the tablet and capsule formulations of paclitaxel following oral administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jackson Christopher, MD, Principal Investigator — Dunedin Hospital
Locations (8):
- Monash Medical Centre, Clayton, Australia
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Dunedin Hospital, Dunedin
  - Wellington Regional Hospital, Wellington
- Taiwan (3):
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Tri-Service General Hospital, Taipei
  - Lotung Poh-Ai Hospital, Yilan
- The Christie NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No